CLINICAL TRIAL: NCT04003506
Title: Comparing the Efficacy of Combining Periarticular Local Infiltration of Analgesia and Adductor Canal Block Using Liposomal Bupivacaine and Standard Bupivacaine in Total Knee Arthroplasty - A Prospective Randomized Controlled Trial
Brief Title: Effectiveness of Adductor Canal Block Using Liposomal Bupivacaine
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Chi-Wing, Consultant, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW19-304
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative
Keywords: bupivacaine; LIA; ACB; total knee replacement; post operative pain; acute pain; anaesthesia
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group LB (Experimental): local infiltration of analgesia (LIA) with adductor canal block (ACB) will be given using 10ml of 1.33% liposomal bupivacaine with 10ml 0.5% standard bupivacaine
  Interventions: Drug: Liposomal bupivacaine
- group SB (Active Comparator): LIA with ACB will be given using 20ml 0.5%standard bupivacaine
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Liposomal bupivacaine — LIA with ACB will be given using 10ml of 1.33% liposomal bupivacaine + 10ml 0.5% standard bupivacaine
  Arms: Group LB
Drug: Bupivacaine Injection — LIA with ACB will be given using 20ml 0.5% standard bupivacaine
  Arms: group SB

SUMMARY:
With aging of population, osteoarthritis of knees and hips become major orthopaedic problems in Hong Kong. Osteoarthritis of knees and hips are associated with significant pain problem and functional disability. Total joints replacement is the ultimate surgical procedures to deal with such problems.

However total joints replacement is associated with significant tissue damage and post-operative pain problems, which would affect post-operative recovery and rehabilitation.

The primary aims of total knee replacement are improvement in functional activities and reduce pain due to degenerated knee joints. However, there are around 20-30% of patients would develop significant pain problem despite uncomplicated total knee replacement. It accounts for major post-operative problems and burdens.

Procedure specific analgesic method with multi-model analgesia technique is well-known to be useful in post-operative pain management, which reduces the post-operative pain score. However, despite using of multi-modal analgesic technique, pain after total joint replacement is still the most unsolved issue. It prolongs the recovery period and increases post-operative analgesic consumptions.

Multimodal analgesia, including periarticular local infiltration of analgesia (LIA), regional nerve block, opioid and non-opioid have been shown to be effective in managing postoperative pain.

Periarticular LIA has been shown to be an effective way of pain management. Regional nerve block using femoral nerve block or adductor canal block (ACB) is also a well-established anlagesic technique after total knee replacement. Comparing with femoral nerve block, it involves more sensory blockade so has the advantage of quadriceps sparing, less affecting the post-operative mobilization.

From most recent systematic reviews and randomized controlled trials, it becomes clear that periarticular LIA has better pain control with less opioid consumption than ACB alone. However, duration of a single-dose LIA may not be long enough after total knee replacement. Recent meta-analysis has shown that combined ACB with LIA could significantly reduce pain scores and morphine consumption compared LIA alone after TKA. Standard bupivacaine, levobupivocaine, ropivocaine were used in ACB in these studies. They are local anaesthetic with half-life ranging from 3-6 hours.

With the availability of liposomal bupivacaine (LB), ACB using LB may further prolong the analgesic effect of ACB as the therapeutic levels of bupivacaine, which are below the toxic range and sustained for 72 hours after injection. Therefore, the issue is whether ACB using LB has even longer analgesic effect than plain bupivacaine or ropivacaine. There was only one study directly compared ACB using LB and 0.1% ropivociane infusion. It was shown that LB had significant impact in pain control in the first 36 hours. However, this was a retrospective study and there was difference in delivery of local anaesthetics (single shot injection for liposomal bupivacaine but continuous infusion for ropivacaine).

The primary aim of this study is to investigate whether ACB using liposomal bupivacaine has even longer analgesic effect than standard bupivacaine (SB) and its cost effectiveness. Secondary aims are to evaluate the pharmacokinetic data of standard bupivacaine and liposomal bupivacaine in adductor canal block and pharmacokinetic data of ropivocaine level in LIA.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-80 years old
* Scheduled for elective primary unilateral total knee replacement
* Chinese patients
* BMI < 40
* Able to speak and understand Cantonese
* Able to provide informed oral and written consent

Exclusion Criteria:

* Revision total knee replacement
* Single stage bilateral total knee replacement
* Known allergy to opioids, local anaesthetic drugs, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDS) including COX-2 inhibitors
* History of chronic pain other than chronic knee pain
* History of immunosuppression
* Daily use of glucocorticoids
* Daily use of strong opioids (morphine, fentanyl, hydromorphone, ketobemidone, methadone, nicomorphine, oxycodone, or meperidine)
* History of severe heart disease (NYHA 2)
* Alcohol or drug abuse
* Impaired renal function, defined as preoperative serum creatinine level over 120 μmol/L
* Pre-existing neurological or muscular disorders
* Psychiatric illness or neurologic or psychiatric diseases potentially influencing pain perception
* Impaired or retarded mental state
* Difficulties in using patient controlled analgesia (PCA)
* Pregnancy
* Local infection
* On immunosuppresants
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pain assessed by numerical rating scales (NRS) pain scores | at postoperative day 1
  NRS pain scores (from 0-10, where 0 is the least satisfaction and 10 most satisfaction) will be recorded during movement and at rest, by NRS (movement) and NRS (rest) respectively

SECONDARY OUTCOMES:
Range of motion (ROM) of knee | from postoperative day 0 until postoperative day 6
  Active and Passive ROM of knee (flexion and extension) will be recorded.
Walking Distance | from postoperative day 0 until postoperative day 6
  Walking distance will be measured in meters
Degree of assistance | from postoperative day 0 until postoperative day 6
  Patients' ability to walk will be assessed. There are three categories including walking without help, walking with walking frame and being unable to walk
Ability to preform straight leg raising | from postoperative day 0 until postoperative day 6
  Patients' ability to preform straight leg raising is recorded after surgery
Plasma level of bupivacaine and ropivacaine. | at before ACB, 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, 16 hours, 20 hours, 24 hours, 48 hours, and 72 hours after ACB.
  Blood sample would be collected and plasma level of bupivacaine and ropivacaine would be measured using liquid chromatography coupled mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Wing Chan, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong